CLINICAL TRIAL: NCT05607381
Title: Neural Mechanisms of Meditation-Based Interventions for Chronic Low Back Pain
Brief Title: Neural Mechanisms of Meditation for Opioid-Treated Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Eric Garland, Associate Dean for Research, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00133405
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain; Opioid Use
MeSH Terms: conditions — Low Back Pain | interventions — Meditation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness (Experimental): A well-validated mindfulness meditation-based therapy [8 sessions] is used to teach patients to independently practice meditation to cope with pain.
  Interventions: Behavioral: Meditation; Other: Usual care
- Meditation (Experimental): A validated meditation-based therapy [8 sessions] is used to teach patients to independently practice meditation to cope with pain.
  Interventions: Behavioral: Meditation; Other: Usual care
- Usual Care (Active Comparator): Patients will receive usual medical care for chronic low back pain.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Meditation — Participants will complete 8 sessions of meditation training with therapy as a means of coping with chronic pain and opioid-related issues.
  Arms: Meditation; Mindfulness
Other: Usual care — Participants will receive usual care for chronic low back pain (e.g., analgesic medication, pain management consultant from a physician, physical therapy, etc.).

SUMMARY:
The purpose of this research study is to see how a mindfulness meditation-based intervention affects pain. Specifically, we are interested in understanding the pain-relieving brain mechanisms of mindfulness meditation-based therapy for patients with opioid-treated chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

1) men/women 18-65 years of age; 2) current chronic low back pain classified according to the NIH Pain Consortium task force research standards for chronic low back pain (pain on at least half the days in the past 6 months); usual back pain ≥3 on 0-10 scale with opioid medication; and 4) current use of prescription opioids for ≥3 months.

Exclusion Criteria:

1) Prior experience with MBSR, MBCT, MORE, or extensive involvement in any standardized meditation training, 2) current cancer diagnosis, 3) suicide intent or attempt in the past 30 days, 4) psychosis or moderate/severe non-opioid substance use disorder in past 6 months; 5) persons with any electronic objects or certain metal objects in their head or body that are incompatible with MRI; 6) those who have had an abnormal brain MRI in the past; 7) those unable to lie still on their back for 1 to 1.5 hours; and 8) pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood oxygenation level dependent (BOLD) signaling | At baseline and at post-treatment (8 weeks)
  Changes in blood oxygenation levels to thermally noxious stimuli (48°C) will be assessed.

SECONDARY OUTCOMES:
Visual Analog Scale Pain Ratings | At baseline and at post-treatment (8 weeks)
  Psychophysical Assessment of Pain: As previously in all of our previous pain studies, pain intensity and unpleasantness ratings will be assessed with a Visual Analog Scale. These scales 1) provide reliably separate assessment of experimental and clinical pain intensity and unpleasantness, 2) are internally consistent, and 3) approximate ratio scale measurement accuracy. The minimum rating ("0") is designated as "no pain" whereas the maximum ("10") is labeled as "most intense imaginable" or "most unpleasant imaginable".
Chronic pain symptoms | At baseline, post-treatment (8 weeks), and 3-month follow-up
  Scores on Brief Pain Inventory, with higher scores indicating higher pain severity (min 0, max 10)
Opioid dose | At baseline, post-treatment (8 weeks), and 3-month follow-up
  Opioid dose as assessed with Timeline Followback Procedure
Pain catastrophizing | At baseline, post-treatment (8 weeks), and 3-month follow-up
  This is a 13-item questionnaire with 3 subscales assessing rumination, magnification, and helplessness in patients. A numeric value between 0 (not at all) and 4 (all the time) is provided in response to each statement. Scores on this assessment range from 0 to 52, with higher values reflecting more salient impacts of pain on one's day to day experience.
Self-transcendence | At baseline, post-treatment (8 weeks), and 3-month follow-up
  Self-transcendence measured by Nondual Awareness Dimensional Assessment, with higher scores indicating higher self-transcendence (min 13, max 65)
Mindful reinterpretation of pain sensations | At baseline, post-treatment (8 weeks), and 3-month follow-up
  Mindful reinterpretation of pain sensations measured by the Mindful Reinterpretation of Pain Sensations Scale, with higher scores indicating higher reinterpretation of pain sensations (min 0, max 45)
Trait mindfulness | At baseline, post-treatment (8 weeks), and 3-month follow-up
  This is a 39-item multidimensional measure of trait mindfulness and includes five subscales: non-reactivity, nonjudgment, describing, observing, and acting with awareness. A numeric value between 1 (never or very rarely true) and 5 (very often or always true) is provided in response to each statement.

OTHER OUTCOMES:
Heart rate variability | At baseline and at post-treatment (8 weeks)
  Changes in heart rate variability (HRV) measured with a 3-lead ECG.
Cue-reactivity | At baseline and at post-treatment (8 weeks)
  Cue-reactivity as evidenced by blood oxygenation level dependent (BOLD) signaling and cue-reactivity ratings during cue-exposure

CONTACTS AND LOCATIONS:
Overall Officials: Eric Garland, PhD, Principal Investigator — University of Utah; Fadel Zeidan, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - Center on Mindfulness and Integrative Health Intervention Development, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The research team will adhere to the NIH Grants Policy on Availability of Research Results: Publications, Intellectual Property Rights, and Sharing Biomedical Research Resources.
Time Frame: Data will become available after the publication of the main study findings from the final data set. Data will be made permanently available.
Access Criteria: Data will be made available upon reasonable request with a signed data access agreement.